CLINICAL TRIAL: NCT03304249
Title: Rural Disparities in Pediatric Obesity: The iAmHealthy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iAmHealthy 2; R01NR016255-01A1 (NIH)
Record Dates: First submitted 2017-09-28; First posted 2017-10-06 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iAmHealthy (Experimental): Participants randomized to this arm receive the iAmHealthy Healthy Lifestyles Program.
  Interventions: Behavioral: iAmHealthy Healthy Lifestyles Program
- Control (Active Comparator): Participants randomized to this group receive comparable content delivered via a newsletter.
  Interventions: Other: Newsletter

INTERVENTIONS:
Behavioral: iAmHealthy Healthy Lifestyles Program — iAmHealthy is behavioral intervention focused on nutrition, behavior and physical activity that engages parents and children in treatment using mobile health (mHealth) technology. Meetings are approximately one hour. Participants will log in for 8 weekly group sessions, followed by 6 monthly sessions.
  Arms: iAmHealthy
Other: Newsletter — Weight loss materials delivered via a newsletter. Each newsletter will cover nutritional, exercise, and behavioral suggestions to improve the child's health. The newsletter will be sent in the mail once a month for 8 months.
  Arms: Control

SUMMARY:
The purpose of this study is to learn if providing a family-based group program using mobile health technology (iAmHealthy Healthy Lifestyles Program) is effective at improving child weight, nutrition, and physical activity.

DETAILED DESCRIPTION:
This is a cluster-randomized study that will test the iAmHealthy Healthy Lifestyles Program versus a standard approach to weight loss in kids current in 2nd thru 4th grade. The iAmHealthy Healthy Lifestyles Program utilizes mobile tools to deliver the weight loss program to kids and families in rural settings. This study will include kids from schools in rural cities/counties, and their parents, and they will be randomly assigned to a group by their school.

The iAmHealthy Healthy Lifestyles Program is a rurally tailored telemedicine intervention. It delivers behavioral, nutritional, and physical activity topics for kids and their families. The total length of the intervention will be about 8 months, which coincides with the length of a typical school year.

ELIGIBILITY:
Inclusion Criteria:

* Family lives in a rural area (city and/or county population less than 20,000)
* Child Body Mass Index (BMI) >85th and <99th percentile
* Child in 2nd thru 4th grade
* Child and Parent speak English
* Family is available at times intervention is offered

Exclusion Criteria:

* Child has physical limitation or receives an injury which significantly limits physical mobility
* Child has significant medical issue
* Child and Parents have significant developmental delay or cognitive impairment
* Child has a sibling who has already enrolled in the program
* Family moves to a non-participating school

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Davis, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Lancaster B, Goldenberg E, Trofimoff AS, Dai Y, Forseth B, Romine RS, Fleming K, Davis A. Mental health outcomes of a pediatric-focused obesity randomized control trial in rural communities. Health Psychol. 2025 Dec;44(12):1095-1104. doi: 10.1037/hea0001518. Epub 2025 May 29. PMID 40440117
- [Derived] Forseth B, Davis AM, Bakula DM, Murray M, Dean K, Swinburne Romine RE, Fleming K. Validation of remote height and weight assessment in a rural randomized clinical trial. BMC Med Res Methodol. 2022 Jul 11;22(1):185. doi: 10.1186/s12874-022-01669-8. PMID 35818033
- [Derived] Davis AM, Beaver G, Dreyer Gillette M, Nelson EL, Fleming K, Swinburne Romine R, Sullivan DK, Lee R, Pettee Gabriel K, Dean K, Murray M, Faith M. iAmHealthy: Rationale, design and application of a family-based mHealth pediatric obesity intervention for rural children. Contemp Clin Trials. 2019 Mar;78:20-26. doi: 10.1016/j.cct.2019.01.001. Epub 2019 Jan 7. PMID 30630108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 18 rural schools between 2017 and 2020.
Pre-assignment Details: Of the 501 children assessed for eligibility, 148 were eligible, consented, and completed baseline measures, each of whom had a parent/caregiver participate with them.
Units Other Than Participants: schools
Period: Overall Study
Arm/Group | iAmHealthy | Control
Started (0 months) | 128; 9 schools (64 pediatric participants and 64 adult participants from 9 schools) | 168; 9 schools (84 pediatric participants and 84 adult participants from 9 schools)
8 Months | 118; 9 schools (59 pediatric participants and 59 adult participants from 9 schools) | 166; 9 schools (83 pediatric participants and 83 adult participants from 9 schools)
Completed (20 months) | 104; 9 schools (52 pediatric participants and 52 adult participants from 9 schools) | 154; 9 schools (77 pediatric participants and 77 adult participants from 9 schools)
Not Completed | 24; 0 schools | 14; 0 schools
Not completed — Lost to Follow-up | 8 | 10
Not completed — Withdrawal by Subject | 12 | 2
Not completed — Moved Out of District | 4 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data collection was focused on child participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | iAmHealthy | Control | Total
Number analyzed (Participants) | 64 | 84 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] — Child age
  years | 8.9880 (0.8859) | 8.8880 (0.8402) | 8.9313 (0.8587)
Sex: Female, Male [Count of Participants; unit: Participants] — Child sex
  Participants
    Female | 38 | 46 | 84
    Male | 26 | 38 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Child ethnicity
  Participants
    Hispanic or Latino | 6 | 14 | 20
    Not Hispanic or Latino | 58 | 70 | 128
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Child race/ethnicity
  Participants
    White | 55 | 74 | 129
    Native American | 0 | 1 | 1
    Asian/Pacific Islander | 1 | 0 | 1
    Other | 1 | 1 | 2
    Biracial | 7 | 8 | 15
Eligible for Free or Reduced Lunch [Count of Participants; unit: Participants]
  Eligible | 36 | 38 | 74
  Not Eligible | 28 | 46 | 74
Approximate Total Household Income (Before Taxes) [Count of Participants; unit: Participants]
  Less than $30,000 | 11 | 24 | 35
  $30,000 to $69,999 | 27 | 25 | 52
  $70,000 to $99,999 | 11 | 25 | 36
  $100,000 to $149,999 | 14 | 7 | 21
  $150,000 or more | 1 | 3 | 4
Body Mass Index Z-Score [Mean (Standard Deviation); unit: z-score] — Body mass index z-score (BMIz) is the age and sex standardized body mass index for children. To calculate BMIz, the equation BMIz = [(BMI/M)^L - 1] ÷ (L × S) is used where M is the median, L is the power transformation to achieve normality, and S is the coefficient of variation. A z-score of 0 represents the historical population norm. A higher BMIz is indicative of higher fat mass. Population: Four participants in the control group did not complete baseline height/weight measurement.
  z-score
    number analyzed (Participants) | 64 | 80 | 144
    (all) | 1.7767 (0.5406) | 1.9209 (0.4705) | 1.8568 (0.5062)
Child's Grade [Count of Participants; unit: Participants]
  2 | 18 | 22 | 40
  3 | 20 | 33 | 53
  4 | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Child Body Mass Index Z-score (BMIz) at Baseline and Month 8
Description: Body mass index z-score (BMIz) is the age and sex standardized body mass index for children. To calculate BMIz, the equation BMIz = [(BMI/M)^L - 1] ÷ (L × S) is used where M is the median, L is the power transformation to achieve normality, and S is the coefficient of variation. A z-score of 0 represents the historical population norm. A higher BMIz is indicative of higher fat mass.
Time Frame: Baseline to Month 8
Population: Six children in the iAmHealthy group and four children in the Control group dropped out or did not complete the height/weight measure at Month 8.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 64 | 80
Z-score
  Baseline | 1.78 (0.54) | 1.92 (0.47)
  Month 8: number analyzed (Participants) | 58 | 76
  Month 8 | 1.78 (0.54) | 1.96 (0.48)

2. Secondary Outcome: Child Body Mass Index Z-score (BMIz) at Baseline and Month 20
Description: as for outcome 1
Time Frame: Baseline to Month 20
Population: Fourteen children in the iAmHealthy group and five children in the Control group dropped out or did not complete the height/weight measure at Month 20.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 64 | 80
Z-score
  Baseline | 1.78 (0.54) | 1.92 (0.47)
  Month 20: number analyzed (Participants) | 50 | 75
  Month 20 | 1.82 (0.50) | 2.04 (0.46)

3. Secondary Outcome: Physical Activity - Average Minutes of Moderate to Vigorous Physical Activity Per Day
Description: Measured using ActiGraph physical activity monitors. Outcome will be calculated as the average (across valid wear days) time spent per day in moderate to vigorous physical activity (MVPA).
Time Frame: Baseline, Month 8, Month 20
Population: Participants dropped out between time points or didn't complete all measures.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 61 | 82
minutes per day
  Baseline | 51.14 (22.72) | 52.95 (18.99)
  Month 8: number analyzed (Participants) | 50 | 66
  Month 8 | 47.16 (18.82) | 49.07 (22.49)
  Month 20: number analyzed (Participants) | 43 | 58
  Month 20 | 44.86 (18.81) | 41.37 (18.57)

4. Secondary Outcome: Physical Activity - % Time in Sedentary Activity
Description: Measured using ActiGraph physical activity monitors. Outcome was calculated as the percentage of time time spent in sedentary activity compared to wear time.
Time Frame: Baseline, Month 8, Month 20
Population: Participants dropped out between time points or didn't complete all measures.
Measure: Mean (Standard Deviation); unit: percent of time sedentary
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 61 | 82
percent of time sedentary
  Baseline | 59.14 (7.12) | 56.57 (6.60)
  Month 8: number analyzed (Participants) | 50 | 66
  Month 8 | 61.14 (8.55) | 59.62 (9.00)
  Month 20: number analyzed (Participants) | 43 | 58
  Month 20 | 63.89 (8.09) | 63.28 (8.11)

5. Secondary Outcome: Photo-assisted 24 Hour Food Recall (24hr FR) - Servings of Fruits and Vegetables
Description: The photo assisted 24hr FR is a standardized five-pass method, developed by the US Department of Agriculture for use in national dietary surveillance.
Time Frame: Baseline, Month 8, Month 20
Population: Participants dropped out between time points or didn't complete all measures.
Measure: Mean (Standard Deviation); unit: servings of fruits and vegetables
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 61 | 80
servings of fruits and vegetables
  Baseline | 3.27 (1.66) | 2.68 (1.38)
  Month 8: number analyzed (Participants) | 48 | 70
  Month 8 | 3.04 (1.68) | 2.45 (1.41)
  Month 20: number analyzed (Participants) | 48 | 68
  Month 20 | 2.89 (1.58) | 2.58 (1.16)

6. Secondary Outcome: Photo-assisted 24 Hour Food Recall (24hr FR) - Servings of Sugar-sweetened Beverages
Description: The photo assisted 24hr FR is a standardized five-pass method, developed by the US Department of Agriculture for use in national dietary surveillance/
Time Frame: Baseline, Month 8, Month 20
Population: Participants dropped out between time points or didn't complete all measures.
Measure: Mean (Standard Deviation); unit: servings of sugar-sweetened beverages
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 61 | 80
servings of sugar-sweetened beverages
  Baseline | 1.19 (0.89) | 1.14 (0.99)
  Month 8: number analyzed (Participants) | 48 | 70
  Month 8 | 0.75 (0.66) | 1.08 (0.89)
  Month 20: number analyzed (Participants) | 48 | 68
  Month 20 | 0.93 (0.84) | 1.21 (1.06)

7. Secondary Outcome: Photo-assisted 24 Hour Food Recall (24hr FR) - Servings of "Red Foods" (Foods High in Sugar and/or Fat)
Description: as for outcome 5
Time Frame: Baseline, Month 8, Month 20
Population: Participants dropped out between time points or didn't complete all measures.
Measure: Mean (Standard Deviation); unit: servings of red foods
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 61 | 80
servings of red foods
  Baseline | 6.64 (2.43) | 7.40 (3.91)
  Month 8: number analyzed (Participants) | 48 | 70
  Month 8 | 5.12 (1.89) | 6.28 (2.28)
  Month 20: number analyzed (Participants) | 48 | 68
  Month 20 | 5.69 (2.00) | 6.89 (2.31)

8. Secondary Outcome: Parent Body Mass Index (BMI)
Description: Parent BMI was calculated at three time points.
Time Frame: Baseline, Month 8, Month 20
Population: Nine parents in the iAmHealthy group and six parents in the Control group dropped out or did not complete the height/weight measure at Month 8. Fourteen parents in the iAmHealthy group and seven parents in the Control group dropped out or did not complete the height/weight measure at Month 20.
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | iAmHealthy | Control
Number analyzed (Participants) | 63 | 80
kg/m²
  Baseline | 35.83 (9.14) | 33.69 (8.81)
  Month 8: number analyzed (Participants) | 54 | 74
  Month 8 | 35.94 (9.73) | 33.79 (9.32)
  Month 20: number analyzed (Participants) | 49 | 73
  Month 20 | 35.23 (9.03) | 34.31 (9.53)

ADVERSE EVENTS:
Time Frame: 20 months
Description: Parents and children were both considered enrolled. No deaths or serious or other adverse events were reported throughout the study.
Arm/Group | iAmHealthy | Control
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/168
Other Adverse Events (participants affected / at risk) | 0/128 | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT03304249/Prot_SAP_000.pdf